CLINICAL TRIAL: NCT06892964
Title: Prospective and Retrospective Clinical Study of Lymphatic Malformations: Institution of an Italian REGistry of Lymphatic Malformations and of a Biobank for Biological Sample Collection
Brief Title: Institution of an Italian Registry and Biobank for Biological Sample Collection
Acronym: IReg-LM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6221
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-07

CONDITIONS: Lymphatic Malformation; Lymphatic Abnormality; Lymphangioma; Lymphatic Abnormalities
MeSH Terms: conditions — Lymphatic Abnormalities; Lymphangioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pstients with isolated lymphatic malformation (Experimental): Genetic profiling (targeted NGS panel) performed on affected tissue sample
  Interventions: Genetic: Genetic profiling of all eligible patients

INTERVENTIONS:
Genetic: Genetic profiling of all eligible patients — Performed genetic profiling in DNA extracted from fresh tissue or FFPE in all patients affected by lymphatic malformation recruited

SUMMARY:
Lymphatic malformations (ML), are benign non-neoplastic, rare, resulting from an embryologic abnormal development of the lymphatic system. Sometimes they may be associated with other vascular malformations (venous or arterial)1,2. ML usually appear at birth, in early childhood or during the first years of life (congenital vs. acquired) and are mainly localized in the region of the head and neck, armpits, groin, retroperitoneal tissues, tongue and mucous membranes of the oral cavity since these areas contain a plethora of lymphatic structures1. The main complications due to their location are airway obstruction, difficulty in eating, and bleeding3-5. Infection and bleeding can promote the sudden, progressive and accelerated growth of these lesions1. The location, speed of growth, and the subsequent complications associated with ML, determine the overall severity of the clinical picture and require generally the referral of the affected patient to a specialized center that can ensure a multidisciplinary care3,5. Recently, the International Society for the Study of Vascular Anomalies (ISSVA), has revised and updated the classification of such malformations, emphasizing the distinction between isolated forms and ML in the context of more complex syndromes with multisystem involvement2. Until a few years ago, the only treatment strategies available for ML were scleroembolization, cryotherapy, transcutaneous laser photocoagulation, and surgical resection of the malformation. The recent identification of genetic alterations in the phosphatidylinositol-3-kinase (PI3K)/protein kinase B (AKT)/target mammalian pathway of rapamycin (mTOR), which underlies many isolated and syndromic ML pictures6-9, has opened up important prospects for personalized treatment with repurposed drugs6,7,10-20. Over the years, the rarity and complexity of ML management have resulted in a fragmented nature of available information and poor nationwide sharing of diagnostic-clinical-assistance-therapeutic protocols (PDTAs) with the consequent need for many families to undertake multispecialty consultations in various provinces or regions before identifying a suitable Referral Center. In addition, recent acquisitions in genetics have forced specialists, a further reevaluation of those complex clinical pictures of ML, whether isolated or syndromic, that could be candidates for personalized drug treatments.

The institution of a national Registry of pathology promoted by the Association of Patients with Lymphatic Malformations, which supports clinicians and families in filling unmet information and clinical care gaps, is a priority project in order to improve the quality of life of patients and the level of care offered to them. In addition, the establishment of a collection of biological specimens, processed according to high quality standards, within a Research Biobank provides the opportunity for patients and their families to maximize the visibility of the specimens, promoting their use in national and international research projects dedicated to ML, in compliance with ELSI (Ethical, Social, and Legal Issues) criteria.

The study primary Objective is To create a computerized registry for ML that collects both retrospective and prospective data in order to estimate the incidence and prevalence of ML, in different phenotypes.

As secondary objectives. (i) Establish a collection of biological specimens (Fresh and fixed biopsy tissue; DNA extracted from whole blood, saliva and where possible from biopsy tissue) within the FPG Research Biobank, intended for future research purposes and available to the entire scientific community; ii) Genetically profile patients who have never undergone molecular diagnostics or who have been tested with restricted panels of genes (PIK3CA, AKT, MTOR, PTEN, KRAS and BRAF) (activity performed on patients per clinical practice); (iii) Define the natural history of ML in different phenotypes and genotypes from prenatal to adult age; (iv) Evaluate the clinical outcomes of different treatments (e.g., experimental drug therapy, maxillofacial surgery, vascular surgery, laser therapy, sclerotherapy, compression therapy, etc.) and different modes of care (type and frequency of visits performed) in the short and long term; (v) Assess the impact of ML on the lives of patients and caregivers; (vi) Support the drafting/updating of national recommendations and standards of care; vii) to promote and facilitate the implementation of research projects dedicated to ML, fostering the advancement of scientific knowledge on this specific disease area;

DETAILED DESCRIPTION:
ENDPOINT Primary endpoint

* To estimate the prevalence and incidence of ML in Italy using data derived from the computerized registry created Secondary endpoints
* To create a collection of biological samples, associated with clinical data, usable by the national and international scientific community (researchers/companies) and aimed at improving knowledge in this field.
* Characterize potential genotype-phenotype associations
* Describe how the phenotype also evolves over time in relation to the genotype found
* Evaluate the short-term (within the first two years after the procedure was performed) and long-term (>2 years) outcome of conservative (vascular laser, scleroembolization, compression therapy), surgical and pharmacological treatment performed by calculating the number of procedures needed during the observation period in the study as well as evaluate the outcome of specialist center intake by calculating the number of patients lost to follow-up, number of patients who changed centers, choice of single-specialty vs multispecialty follow-up;
* Analyze responses to questionnaires on quality of life, pain, sleep quality, adaptive skills, and parenting stress;
* Define a nationally shared diagnostic for ML.

References:

1. https://snlg.iss.it/wp-content/uploads/2021/04/LG-276-Anomalie-Vascolari.pdf
2. International Society for the Study of Vascular Anomalies. ISSVA Classification of Vascular Anomalies ©. Published 2018. Accessed May 13, 2022. issva.org/classification
3. Leboulanger N, Bisdorff A, Boccara O, Dompmartin A, Guibaud L, Labreze C, Lagier J, Lebrun- Vignes B, Herbreteau D, Joly A, Malloizel-Delaunay J, Martel A, Munck S, Saint-Aubin F, Maruani A. French national diagnosis and care protocol (PNDS, protocole national de diagnostic et de soins): cystic lymphatic malformations. Orphanet J Rare Dis. 2023 Jan 13;18(1):10. doi: 10.1186/s13023- 022-02608-y
4. Ghaffarpour N, Baselga E, Boon LM, Diociaiuti A, Dompmartin A, Dvorakova V, El Hachem M, Gasparella P, Haxhija E, Kyrklund K, Irvine AD, Kapp FG, Rößler J, Salminen P, van den Bosch C, van der Vleuten C, Kool LS, Vikkula M. The VASCERN-VASCA working group diagnostic and management pathways for lymphatic malformations. Eur J Med Genet. 2022 Dec;65(12):104637. doi: 10.1016/j.ejmg.2022.104637. Epub 2022 Oct 9. PMID: 36223836.
5. Moneghini L, Sangiorgio V, Tosi D, Colletti G, Melchiorre F, Baraldini V, Graziani D, Alfano RM, Vercellio G, Bulfamante G. Head and neck vascular anomalies. A multidisciplinary approach and diagnostic criteria. Pathologica. 2017 Mar;109(1):47-59. PMID: 28635993.
6. Lee SY, Loll EG, Hassan AES, Cheng M, Wang A, Farmer DL. Genetic and Molecular Determinants of Lymphatic Malformations: Potential Targets for Therapy. J Dev Biol. 2022;10(1). doi:10.3390/jdb10010011
7. Snyder E, Sarma A, Borst AJ, Tekes A. Lymphatic Anomalies in Children: Update on Imaging Diagnosis, Genetics and Treatment. Am J Roentgenol. Published online 2022. doi:10.2214/ajr.21.27200
8. Nathan N, Keppler-Noreuil KM, Biesecker LG, Moss J, Darling TN. Mosaic Disorders of the PI3K/PTEN/AKT/TSC/mTORC1 Signaling Pathway. Dermatol Clin. 2017;35(1):51-60. doi:10.1016/j.det.2016.07.001
9. Gomes IP, Guimarães LM, Pereira T dos SF, et al. Assessment of PI3K/AKT and MAPK/ERK pathways activation in oral lymphatic malformations. Oral Surg Oral Med Oral Pathol Oral Radiol. 2022;133(2):216-220. doi:10.1016/j.oooo.2021.08.018
10. Wu C, Song D, Guo L, Wang L. Refractory Head and Neck Lymphatic Malformation in Infants Treated With Sirolimus: A Case Series. Front Oncol. 2021;11:616702. doi:10.3389/fonc.2021.616702
11. Holm A, Te Loo M, Schultze Kool L, et al. Efficacy of Sirolimus in Patients Requiring Tracheostomy for Life-Threatening Lymphatic Malformation of the Head and Neck: A Report From the European Reference Network. Front Pediatr. 2021;9:697960. doi:10.3389/fped.2021.697960
12. Amodeo I, Colnaghi M, Raffaeli G, et al. The use of sirolimus in the treatment of giant cystic lymphangioma: Four case reports and update of medical therapy. Medicine (Baltimore). 2017;96(51):e8871. doi:10.1097/MD.0000000000008871
13. Holm A, Te Loo M, Schultze Kool L, et al. Efficacy of Sirolimus in Patients Requiring Tracheostomy for Life-Threatening Lymphatic Malformation of the Head and Neck: A Report From the European Reference Network. Front Pediatr. 2021;9:697960. doi:10.3389/fped.2021.697960
14. Amodeo I, Colnaghi M, Raffaeli G, et al. The use of sirolimus in the treatment of giant cystic lymphangioma: Four case reports and update of medical therapy. Medicine (Baltimore). 2017;96(51):e8871. doi:10.1097/MD.0000000000008871
15. Ozeki M, Nozawa A, Yasue S, et al. The impact of sirolimus therapy on lesion size, clinical

    symptoms, and quality of life of patients with lymphatic anomalies. Orphanet J Rare Dis. 2019;14(1):141. doi:10.1186/s13023-019-1118-1
16. Triana P, Miguel M, Díaz M, Cabrera M, López Gutiérrez JC. Oral Sirolimus: An Option in the Management of Neonates with Life-Threatening Upper Airway Lymphatic Malformations. Lymphat Res Biol. 2019;17(5):504-511. doi:10.1089/lrb.2018.0068
17. Curry S, Logeman A, Jones D. Sirolimus: A Successful Medical Treatment for Head and Neck Lymphatic Malformations. Case Rep Otolaryngol. 2019;2019:2076798. doi:10.1155/2019/2076798
18. Wenger TL, Ganti S, Bull C, Lutsky E, Bennett JT, Zenner K, Jensen DM, Dmyterko V, Mercan E, Shivaram GM, Friedman SD, Bindschadler M, Drusin M, Perkins JN, Kong A, Bly RA, Dahl JP, Bonilla- Velez J, Perkins JA. Alpelisib for the treatment of PIK3CA-related head and neck lymphatic malformations and overgrowth. Genet Med. 2022 Nov;24(11):2318-2328. doi: 10.1016/j.gim.2022.07.026
19. Shaheen MF, Tse JY, Sokol ES, Masterson M, Bansal P, Rabinowitz I, Tarleton CA, Dobroff AS, Smith TL, Bocklage TJ, Mannakee BK, Gutenkunst RN, Bischoff J, Ness SA, Riedlinger GM, Groisberg R, Pasqualini R, Ganesan S, Arap W. Genomic landscape of lymphatic malformations: a case series and response to the PI3Kα inhibitor alpelisib in an N-of-1 clinical trial. Elife. 2022 Jul 5;11:e74510. doi: 10.7554/eLife.74510. PMID: 35787784; PMCID: PMC9255965.
20. Delestre F, Venot Q, Bayard C, Fraissenon A, Ladraa S, Hoguin C, Chapelle C, Yamaguchi J, Cassaca R, Zerbib L, Magassa S, Morin G, Asnafi V, Villarese P, Kaltenbach S, Fraitag S, Duong JP, Broissand C, Boccara O, Soupre V, Bonnotte B, Chopinet C, Mirault T, Legendre C, Guibaud L, Canaud G. Alpelisib administration reduced lymphatic malformations in a mouse model and in patients. Sci Transl Med. 2021 Oct 6;13(614):eabg0809. doi: 10.1126/scitranslmed.abg0809

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-100 years
2. Signed informed consent.
3. Individuals with any type of ML (isolated, syndromic, congenital or acquired, with or without molecular confirmation) identified by participating centers

Exclusion Criteria:

* Patients whose clinical picture is not compatible with points a) (b) and (c) of the inclusion criteria, as assessed by the Investigator.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2043-06-27 (Estimated); Study Completion 2044-06-27 (Estimated)

PRIMARY OUTCOMES:
Estimate the prevalence and incidence of ML in Italy | 20 years
  Data collection derived from the computerized registry created for the study

SECONDARY OUTCOMES:
Institution of a biobank collecting biological samples of lymphatic malformations | 20 years
  collection of biological samples (blood, buccal swab, tissue), associated with clinical data, usable by the national and international scientific community (researchers/companies) and aimed at improving knowledge in this field.
Characterize potential genotype-phenotype associations | 20years
  The registry institution and the prospective collection of genetic data will allow the definition of potential genotype phenotype association
Natural evolution of lymphatic malformations | 20years
  Describe natural evolution of lymphatic malformations according to genetic defects
Evaluate the short and long-term (< or > 2 years) outcome of LM patients | 20years
  Comparison between of conservative (vascular laser, scleroembolization, compression therapy), surgical and pharmacological treatment performed by calculating the number of procedures needed during the observation period in the study as well as evaluate the outcome of specialist center intake by calculating the number of patients lost to follow-up, number of patients who changed centers, choice of single-specialty vs multispecialty follow-up
Evaluate quality of life status in this specific patient cohort | 20years
  Analyze responses to questionnaires on quality of life, pain, sleep quality, adaptive skills, and parenting stress

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Leoni, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Department of Woman and Child Health and Public Health, Fondazione Policlinico A. Gemelli, IRCCS, Roma, Italy

REFERENCES:
- [Result] Trevisan V, De Corso E, Viscogliosi G, Onesimo R, Cina A, Panfili M, Perri L, Agazzi C, Giorgio V, Rigante D, Vento G, Papacci P, Paradiso FV, Silvaroli S, Nanni L, Resta N, Castori M, Galli J, Paludetti G, Zampino G, Leoni C. A multi-step approach to overcome challenges in the management of head and neck lymphatic malformations, and response to treatment. Orphanet J Rare Dis. 2024 Jul 23;19(1):276. doi: 10.1186/s13023-024-03200-2. PMID 39044220